CLINICAL TRIAL: NCT04597528
Title: Maternal and Perinatal Outcome After Elective Induction of Labour at Thirty Nine Weeks and Zero Days Upto Thirty Nine Weeks and Six Days in Nulliparous Singleton Pregnancies :a Prospective Observational Study in a Tertiary Care Centre
Brief Title: Elective Induction of Labour at Thirty Nine Weeks: a Prospective Observational Study
Acronym: EIOL39
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Athulya Shajan, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 42/19/IEC/JMMC&RI; U1111-1245-7675 (Other: WHO)
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Related
Keywords: Elective induction of labour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective induction group: Nulliparous singleton gestations undergoing elective induction between 39weeks and 0days -39weeks and 6 days based on clinical information and evaluation of the earliest ultrasound as described in Gestational Age
  Interventions: Other: Elective Induction

INTERVENTIONS:
Other: Elective Induction — All patients admitted to the labour room would be approached to be enrolled in the study.
  Those satisfying the inclusion and exclusion criteria would be prospectively enrolled to the study after procuring an informed consent. If a patient appears to meet the criteria for the study, she will be told about the study and asked for written informed consent to participate. Consent may be obtained anytime from 34 weeks 0 days to 38 weeks 6 days of gestation. Data would be procured on a pre set proforma, entered in real time and safely stored.
  The data would later be abstracted to an excel sheet.

SUMMARY:
Adverse events are considered to increase in pregnancies extending beyond 39 weeks.

For multiparous patients, especially those with a favourable cervix, it is perhaps easy to justify an elective induction at 39 weeks given the low risk of caesarean section.

However, for nulliparous patients the current evidence, derived mainly from retrospective observational studies, does not allow a clear recommendation with the exception perhaps of the recent A Randomized Trial of Induction Versus Expectant Management (ARRIVE) trial. Given the reported increased risks of adverse events in pregnancies extending beyond 39 weeks it has been hypothesized that a policy of planned elective induction at 39 weeks could improve outcomes for the infant and the mother. There is a trend towards an increased rate of elective labour induction in pregnancies at 39 weeks, indicating that practitioners are more commonly using elective induction at this gestational age. The practice in India varies slightly from institute to institute.

The investigator intend to study the maternal and perinatal outcome, after elective induction of labour, at thirty nine weeks and zero days upto thirty nine and six days, amongst nulliparous singleton pregnancies followed up for the duration of their hospital stay, in Jubilee Mission Medical College and Research Institute (JMMC and RI).

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous - no previous pregnancy beyond 20 weeks
2. Singleton gestation.
3. Undergoing elective induction between 39weeks and 0days -39weeks and 6 days based on clinical information and evaluation of the earliest ultrasound as described in Gestational Age
4. Consenting to be part of the study

Exclusion Criteria:

1. Plan for caesarean delivery or any contraindication to vaginal delivery
2. Foetal demise or known major foetal anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Singleton nulliparous gestation undergoing elective induction between 39weeks and 0days -39weeks and 6 days
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Caesarean Section (CS) | Till discharge from hospital or upto 4 days from day of delivery whichever is later
  Number of participants who underwent CS measured in percentage
Number of neonates requiring intensive care | 24 hours from birth
  Incidence of admission to neonatal intensive care unit (NICU) requiring cardio respiratory support within the first 24 hours of birth.
  Cardio respiratory support defined as needing any of the following within the first 24 hours of birth
  1. Cardiopulmonary resuscitation (CPR)
  2. invasive mechanical ventilatory care with a definitive airway
  3. high flow nasal cannula (HFNC)
  4. nasal continuous positive airway pressure (CPAP)ventilation

SECONDARY OUTCOMES:
Time to delivery (induction to delivery time ) | 24 hours
  Time taken from induction of delivery to delivery of the baby measured in hours and minutes
Number of study participants with chorioamnionitis | Diagnosed at anytime, through delivery, upto 24 hours after birth
  Chorioamnionitis, documented as a clinical diagnosis before delivery
Number of participants with Postpartum hemorrhage | Upto 12 weeks from day of delivery
  Postpartum hemorrhage, defined as answering "yes" for any of the questions as per a predefined checklist for
Neonatal Mortality | Antepartum upto 30 days post delivery
  Number of neonatal deaths
APGAR</= 7 at birth | Upto 5 mins after birth
  The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Number of infants with meconium aspiration syndrome (MAS) | Delivery through discharge or upto 4 days post delivery whichever is earlier
  Number of infants with MAS

CONTACTS AND LOCATIONS:
Overall Officials: Sareena Gilvaz, MD, DGO, Study Director — Jubilee Mission Medical College and Research Institute; Bindu Menon, MS, Study Chair — Jubilee Mission Medical College and Research Institute; Athulya Shajan, MBBS, Principal Investigator — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India